CLINICAL TRIAL: NCT04365608
Title: Safety and Efficacy of Endotracheal Intubation by Paramedics in Suspected/Confirmed COVID-19 Patients Under Cardiac Arrest Using Vie Scope Laryngoscope
Brief Title: Prehospital Intubation of COVID-19 Patient With Personal Protective Equipment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lazarski University (Other)
Collaborators: Poznan University of Medical Sciences (Other); Wroclaw Medical University (Other); Medical University of Bialystok (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Assoc Prof PhD, Lazarski University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INT_EMS_PPE_1
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Intubation Complication; Intubation; Difficult or Failed; Cardiac Arrest; Influenza; Safety Issues
Keywords: endotracheal intubation; cardiac arrest; personal protective equipment; laryngoscope; Vie Scope; COVID-19; SARS-CoV-2; emergency medicine
MeSH Terms: conditions — Heart Arrest; Influenza, Human; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct laryngoscopy (Active Comparator): Intubation will be done using direct laryngoscopy. The standard intubation procedure is to use a styletted tube and no sedation. When standard laryngoscopy-assisted intubation is not possible, an alternate procedure will be used based on the guidelines on difficult airway management.
  Interventions: Procedure: Direct laryngoscopy
- Vie Scope laryngoscopy (Active Comparator): Intubation will be done using Vie Scope laryngoscopy
  Interventions: Procedure: Vie Scope laryngoscopy

INTERVENTIONS:
Procedure: Direct laryngoscopy — standard laryngoscope with Macintosh blade
  Other Names: MAC
  Arms: Direct laryngoscopy
Procedure: Vie Scope laryngoscopy — Vie Scope with dedicated bougie stylet
  Other Names: VCE
  Arms: Vie Scope laryngoscopy

SUMMARY:
The safety and efficacy of a laryngoscopy as a primary intubation tool in urgent endotracheal intubation of cardiac arrest patients with suspected/confirmed COVID-19 has not been well-described in the literature. This study will answer whether using a Vie Scope laryngoscope will impact on the efficacy and safety of intubation compared with a traditional direct laryngoscopy.

DETAILED DESCRIPTION:
Intubation will be carried out in full personal protective equipment conditions of the operator

ELIGIBILITY:
Inclusion Criteria:

* All adult patients requiring out-of-hospital intubation

Exclusion Criteria:

* Patient under 18 years old
* Patients with criteria predictive of impossible intubation under direct laryngoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Intubation success rate during at the first laryngoscopy | 10 min
  Definition of failed intubation: Time to intubation is longer than 120 seconds or wrong placement of endotracheal tube (For example : Esophageal intubation etc.)

SECONDARY OUTCOMES:
Intubation difficulty Scale score | 10 min
  Intubation difficulty assessed by Intubation difficulty Scale score
Complications related to tracheal intubation | 10 min
  Complications related to tracheal intubation during advanced Cardiopulmonary Resuscitation (CPR): failure, esophageal intubation, mainstem intubation, vomiting, pulmonary aspiration, dental trauma, extubation
Time to completion of tracheal intubation (TI) procedure | 10 min
  Time to completion of tracheal intubation (TI) procedure measured from the instant that the laryngoscope blade touches the patient to the moment that the tracheal tube cuff is inflated
Duration of the interruption of chest compression during ETI procedure | 10 min
  Duration of the interruption of chest compression during ETI procedure
Laryngeal View during intubation | 10 min
  We will record the best laryngeal View during intubation. We will record according to the Cormack-Lehane Grade system.
POGO score | 10 min
  self-reported percentage of glottis opening (POGO) score

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Emergency Medical Service, Poznan
  - Emergency Medical Service, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: after manuscript publishing

REFERENCES:
- [Derived] Szarpak L, Peacock FW, Rafique Z, Ladny JR, Nadolny K, Malysz M, Dabrowski M, Chirico F, Smereka J. Comparison of Vie Scope(R) and Macintosh laryngoscopes for intubation during resuscitation by paramedics wearing personal protective equipment. Am J Emerg Med. 2022 Mar;53:122-126. doi: 10.1016/j.ajem.2021.12.069. Epub 2022 Jan 4. PMID 35016094